CLINICAL TRIAL: NCT02630069
Title: Cytidine-5'-Diphosphate-choline Treatment in Amphetamine Type Stimulant-using Adolescents
Brief Title: CDP-choline Treatment in ATS Users
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, Sujung Yoon, Professor, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIH_ATS
Record Dates: First submitted 2015-12-06; First posted 2015-12-15 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Substance Use Disorders
Keywords: amphetamine type stimulant; adolescents
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CDP-choline+supportive psychotherapy (Experimental): CDP-choline 500mg once a day for 12 weeks / Supportive psychotherapy 1 session/2 weeks for 12 weeks
  Interventions: Drug: CDP-choline; Behavioral: Supportive psychotherapy
- Placebo+supportive psychotherapy (Placebo Comparator): Placebo 500mg once a day for 12 weeks / Supportive psychotherapy 1 session/2 weeks for 12 weeks
  Interventions: Drug: Placebo; Behavioral: Supportive psychotherapy
- Healthy control (No Intervention): No intervention

INTERVENTIONS:
Drug: CDP-choline — CDP-choline 500mg once a day for 12 weeks
  Arms: CDP-choline+supportive psychotherapy
Drug: Placebo — Placebo 500mg once a day for 12 weeks
  Arms: Placebo+supportive psychotherapy
Behavioral: Supportive psychotherapy — Supportive psychotherapy 1 session/2 weeks for 12 weeks
  Arms: CDP-choline+supportive psychotherapy; Placebo+supportive psychotherapy

SUMMARY:
This study is a 12-week, randomized, double-blind, placebo-controlled trial of cytidine-5'-diphosphate choline in amphetamine-type stimulants-using adolescents.

DETAILED DESCRIPTION:
This study is a 12-week, randomized, double-blind, placebo-controlled trial of cytidine-5'-diphosphate choline (CDP-choline) in amphetamine-type stimulants-using adolescents. Multi-level assessments will be performed to determine whether CDP-choline administration with supportive psychotherapy, compared to placebo administration with supportive psychotherapy, will 1) repair ATS-induced neural cell damage of the target brain regions, 2) improve cognitive deficits and normalize the relevant target neural circuits, and then 3) reduce ATS-taking behaviors in ATS-using adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14-40 years
* Amphetamine (or amphetamine-like) use disorder (DSM-IV-TR)
* Informed consent
* Seeking treatment

Exclusion Criteria:

* Major medical or neurological illnesses
* Psychiatric illnesses requiring hospitalization, prescription of psychotropic medications, or emergency psychiatric interventions
* Current and past diagnosis of a psychotic disorder, bipolar disorder, conduct disorder, or attention-deficit hyperactivity disorder
* Occasional ATS use (less than monthly use)
* IQ of 80 or lower
* Pregnancy or breastfeeding
* Clinically significant suicidal or homicidal ideation
* Substance use disorders (substances other than amphetamine or MA)

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
the total number of amphetamine- and methamphetamine(MA)-negative samples using urine screening | baseline through 12 weeks
abstinence which is defined as five or more consecutive weeks of amphetamine- and MA-negative samples | baseline through 12 weeks
treatment program retention | baseline through 12 weeks

SECONDARY OUTCOMES:
standardized scores on a neuropsychological test battery | baseline and 12 weeks
number of participants with adverse events | baseline through 12 weeks
structural brain changes in magnetic resonance imaging assessed by computational approaches | baseline and 12 weeks
functional brain changes in magnetic resonance imaging assessed by computational approaches | baseline and 12 weeks
metabolic brain changes in magnetic resonance imaging assessed by computational approaches | baseline and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea